CLINICAL TRIAL: NCT02752828
Title: A Randomized, Active-controlled, Open Label, 2-treatment Arm, and Multicenter Study Comparing the Efficacy and Safety of the Insulin Glargine/Lixisenatide Combination to Insulin Glargine on Top of OADs in Japanese Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination (LixiLan) to Insulin Glargine Alone on Top of Oral Anti-diabetic Drugs (OADs) With Type 2 Diabetes in Japan
Acronym: LIXILAN JP-O2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14114; U1111-1176-8450 (Other: UTN)
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LixiLan (Experimental): LixiLan (insulin glargine/lixisenatide) is injected subcutaneously (under the skin) once daily. Dose is individually adjusted.
  Background therapy with OADs (except dipeptidyl-peptidase-4 inhibitor) should be continued during the treatment period.
  Interventions: Drug: Insulin glargine/lixisenatide (HOE901/AVE0010); Drug: Oral anti-diabetic drugs
- insulin glargine (Active Comparator): Insulin glargine (HOE901) is injected subcutaneously (under the skin) once daily. Dose is individually adjusted.
  Background therapy with OADs (except dipeptidyl-peptidase-4 inhibitor) should be continued during the treatment period.
  Interventions: Drug: Insulin glargine (HOE901); Drug: Oral anti-diabetic drugs

INTERVENTIONS:
Drug: Insulin glargine/lixisenatide (HOE901/AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: LixiLan
  Arms: LixiLan
Drug: Insulin glargine (HOE901) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: insulin glargine
Drug: Oral anti-diabetic drugs — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To compare LixiLan to insulin glargine in glycated hemoglobin (HbA1c) change from baseline to Week 26 in patients with type 2 Diabetes.

Secondary Objective:

To compare the overall efficacy and safety of LixiLan to insulin glargine (with or without OADs) over a 26 Week treatment period in patients with type 2 Diabetes.

DETAILED DESCRIPTION:
The maximum study duration per patient will be approximately 29 weeks: an up to 2-week screening period, a 26-week randomized open-label treatment period and a 3-day post-treatment safety follow up period.

ELIGIBILITY:
Inclusion criteria :

* Patient with type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year before the screening visit, receiving 1 or 2 OADs that can be Biguanide,Thiazolidinedione (TZD), -Alpha-glucosidase-inhibitor (alpha-GI),Sodium glucose co-transporter 2 (SGLT2) inhibitor,Sulfonylurea (SU),Rapid-acting insulin secretagogue (Glinide),diphenyl-peptidase -4 inhibitor (DPP-4 inhibitor).
* Signed written informed consent.

Exclusion criteria:

* At the screening visit: Age <20 years.
* At the screening visit: HbA1c <7.5% or >9.5%.
* At the screening visit: fasting plasma glucose (FPG) >180 mg/dL (10.0 mmol/L).
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Use of oral or injectable glucose-lowering agents other than those stated during the inclusion criteria in the 3 months before the screening visit.
* Previous treatment with insulin (except for short-term treatment due to intercurrent illness including gestational diabetes at the discretion of the trial physician).
* Laboratory findings at the time of screening:
* Amylase and/or lipase: >3 times the upper limit of the normal (ULN) laboratory range,
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST): >3 ULN,
* Calcitonin ≥20 pg/mL (5.9 pmol/L),
* Positive serum pregnancy test in female of childbearing potential.
* Contraindication to use of lixisenatide according to the local labeling. History of hypersensitivity to any Glucagon-Like Peptide-1 Receptor Agonists or to metacresol.
* Contraindication to use of insulin glargine according to local labeling. History of hypersensitivity to insulin glargine or to any of the excipients.
* Patient who has a severe renal function impairment with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 or end-stage renal disease for patient not treated with metformin.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (eg, multiple endocrine neoplasia syndromes).
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy, stomach/gastric surgery.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2016-05-23; Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, 26 weeks

SECONDARY OUTCOMES:
Percentage of patients reaching HbA1c <7% or ≤6.5% | 26 weeks
Change from baseline in 2-hour postprandial glucose (PPG) during standardized meal test | Baseline, 26 weeks
Change from baseline in 7 point self monitored plasma glucose (SMPG) profiles during standardized meal test | Baseline, 26 weeks
Change from baseline in body weight | Baseline, 26 weeks
Percentage of patients reaching HbA1c <7% with no body weight gain and with no documented (PG ≤70 mg/dL [3.9 mmol/L]) symptomatic hypoglycemia | 26 weeks
Percentage of patients reaching HbA1c <7% at Week 26 with no documented (PG ≤70 mg/dL [3.9 mmol/L]) symptomatic hypoglycemia | 26 weeks
Percentage of patients requiring a rescue therapy | 26 weeks
Number of adverse events | 26 weeks
Number of hypoglycemic events | 26 weeks
Measurement of anti-lixisenatide antibodies from baseline | Baseline, 26 weeks
Measurement of anti-insulin antibodies from baseline | Baseline, 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (113):
- Japan (113):
  - Investigational Site Number 392002, Adachi-Ku
  - Investigational Site Number 392132, Annaka-Shi
  - Investigational Site Number 392009, Arakawa-Ku
  - Investigational Site Number 392025, Atsugi-Shi
  - Investigational Site Number 392024, Chiba
  - Investigational Site Number 392151, Chiba
  - Investigational Site Number 392011, Chigasaki-Shi
  - Investigational Site Number 392013, Chiyoda-Ku
  - Investigational Site Number 392052, Chiyoda-Ku
  - Investigational Site Number 392003, Chūōku
  - Investigational Site Number 392017, Chūōku
  - Investigational Site Number 392055, Chūōku
  - Investigational Site Number 392155, Chūōku
  - Investigational Site Number 392008, Fujimi-Shi
  - Investigational Site Number 392143, Fujisawa-Shi
  - Investigational Site Number 392054, Fukuoka
  - Investigational Site Number 392094, Fukuoka
  - Investigational Site Number 392147, Fukuoka
  - Investigational Site Number 392100, Gifu
  - Investigational Site Number 392059, Hachioji-Shi
  - Investigational Site Number 392083, Hakodate-Shi
  - Investigational Site Number 392048, Hamamatsu
  - Investigational Site Number 392102, Hamamatsu
  - Investigational Site Number 392079, Hiki-Gun
  - Investigational Site Number 392112, Hirosaki-Shi
  - Investigational Site Number 392109, Hofu-Shi
  - Investigational Site Number 392057, Iruma-Shi
  - Investigational Site Number 392022, Ise-Shi
  - Investigational Site Number 392020, Izumisano
  - Investigational Site Number 392139, Kagoshima
  - Investigational Site Number 392136, Kamogawa-Shi
  - Investigational Site Number 392066, Kashiwa-Shi
  - Investigational Site Number 392045, Kashiwara-Shi
  - Investigational Site Number 392006, Kasugai-Shi
  - Investigational Site Number 392053, Kawagoe-Shi
  - Investigational Site Number 392065, Kawagoe-Shi
  - Investigational Site Number 392007, Kawaguchi-Shi
  - Investigational Site Number 392062, Kawaguchi-Shi
  - Investigational Site Number 392077, Kawasaki-Shi
  - Investigational Site Number 392082, Kawasaki-Shi
  - Investigational Site Number 392091, Kawasaki-Shi
  - Investigational Site Number 392142, Kawasaki-Shi
  - Investigational Site Number 392133, Kitaazumi-Gun
  - Investigational Site Number 392129, Kitakyushu-Shi
  - Investigational Site Number 392041, Kitakyusyu-Shi
  - Investigational Site Number 392068, Kitakyusyu-Shi
  - Investigational Site Number 392114, Kitamoto-Shi
  - Investigational Site Number 392086, Kobe
  - Investigational Site Number 392044, Koga-Shi
  - Investigational Site Number 392119, Kokubunji-Shi
  - Investigational Site Number 392001, Koriyama-Shi
  - Investigational Site Number 392028, Kumamoto
  - Investigational Site Number 392092, Kumamoto
  - Investigational Site Number 392108, Kumamoto
  - Investigational Site Number 392075, Kure-Shi
  - Investigational Site Number 392032, Kurume-Shi
  - Investigational Site Number 392118, Kushiro
  - Investigational Site Number 392107, Kyoto
  - Investigational Site Number 392088, Maebashi
  - Investigational Site Number 392113, Matsumoto-Shi
  - Investigational Site Number 392122, Minatoku
  - Investigational Site Number 392076, Misato-Shi
  - Investigational Site Number 392042, Mito
  - Investigational Site Number 392078, Mito
  - Investigational Site Number 392148, Nagano
  - Investigational Site Number 392026, Nagoya
  - Investigational Site Number 392101, Nagoya
  - Investigational Site Number 392128, Nagoya
  - Investigational Site Number 392131, Nagoya
  - Investigational Site Number 392134, Nagoya
  - Investigational Site Number 392154, Naka
  - Investigational Site Number 392127, Niigata
  - Investigational Site Number 392050, Niihama-Shi
  - Investigational Site Number 392115, Ogawa-Machi, Hikigun
  - Investigational Site Number 392071, Okayama
  - Investigational Site Number 392095, Onga-Gun
  - Investigational Site Number 392117, Osaka
  - Investigational Site Number 392144, Osaka
  - Investigational Site Number 392040, Oyama-Shi
  - Investigational Site Number 392084, Saga
  - Investigational Site Number 392069, Saijo-Shi
  - Investigational Site Number 392030, Saitama-Shi
  - Investigational Site Number 392074, Sanda-Shi
  - Investigational Site Number 392047, Sapporo
  - Investigational Site Number 392089, Sapporo
  - Investigational Site Number 392150, Sapporo
  - Investigational Site Number 392097, Sasebo-Shi
  - Investigational Site Number 392004, Sendai
  - Investigational Site Number 392103, Sendai
  - Investigational Site Number 392070, Shimonoseki-Shi
  - Investigational Site Number 392034, Shimotsuke-Shi
  - Investigational Site Number 392110, Shinagawa-Ku
  - Investigational Site Number 392021, Shinjuku-Ku
  - Investigational Site Number 392098, Shinjuku-Ku
  - Investigational Site Number 392037, Shizuoka
  - Investigational Site Number 392081, Shizuoka
  - Investigational Site Number 392019, Shobara-Shi
  - Investigational Site Number 392018, Shunan-Shi
  - Investigational Site Number 392027, Suita-Shi
  - Investigational Site Number 392056, Taito-Ku
  - Investigational Site Number 392146, Takamatsu
  - Investigational Site Number 392051, Takatsuki-Shi
  - Investigational Site Number 392061, Tokorozawa-Shi
  - Investigational Site Number 392111, Tomakomai-Shi
  - Investigational Site Number 392029, Toyonaka-Shi
  - Investigational Site Number 392073, Tsu
  - Investigational Site Number 392063, Ube-Shi
  - Investigational Site Number 392093, Ube-Shi
  - Investigational Site Number 392039, Yamato-Shi
  - Investigational Site Number 392067, Yatsushiro-Shi
  - Investigational Site Number 392012, Yokohama
  - Investigational Site Number 392126, Yokohama
  - Investigational Site Number 392035, Zentsuji-Shi

REFERENCES:
- [Result] Terauchi Y, Nakama T, Spranger R, Amano A, Inoue T, Niemoeller E. Efficacy and safety of insulin glargine/lixisenatide fixed-ratio combination (iGlarLixi 1:1) in Japanese patients with type 2 diabetes mellitus inadequately controlled on oral antidiabetic drugs: A randomized, 26-week, open-label, multicentre study: The LixiLan JP-O2 randomized clinical trial. Diabetes Obes Metab. 2020 Sep;22 Suppl 4:14-23. doi: 10.1111/dom.14036. PMID 32291880